CLINICAL TRIAL: NCT02603900
Title: A Double-Blinded Randomized Controlled Trial Comparing the Adductor Canal Catheter (ACC) and Local Infiltration of Analgesia (LIA) Following Primary Total Knee Arthroplasty
Brief Title: Adductor Canal Catheter vs Local Infiltration of Analgesia for Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Jaime Baratta, Assistant Professor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15D.490
Record Dates: First submitted 2015-10-22; First posted 2015-11-13 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Acute Pain; Regional Anesthesia Morbidity
Keywords: Adductor Canal Catheter; Arthroplasty, Replacement, Knee; Local infiltration of analgesia
MeSH Terms: conditions — Acute Pain | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor Canal Catheter (Experimental): This group will receive ropivacaine 0.5% 15 ml for the adductor canal block under ultrasound guided nerve block. A multi-orifice catheter will be placed in the adductor canal and an infusion of ropivacaine 0.2% at 10 ml/hr will be continued for 72 hours.
  Interventions: Drug: ropivacaine; Device: Adductor Canal Catheter
- Local Infiltration of Analgesia (Experimental): Local infiltration using 20 ml of free bupivacaine solution (Marcaine 0.25% with epinephrine 1:200000, ) diluted with 40 ml of normal saline following implantation of the knee prosthesis, the solution will be injected into the vastus medialis (5 ml), medial retinaculum (5 ml), origin of MCL (5 ml) and LCL (5 ml), lateral portion of quadriceps tendon (5 ml), vastus lateralis (5 ml), and subcutaneous tissues especially along saphenous nerve distribution (30 ml). Postoperatively, a sham adductor canal catheter will be placed as in the ACC arm following stabilization in the PACU to infuse only normal saline with an initial bolus of 15 ml saline and infusion of saline at 10ml/hr for 72 hours.
  Interventions: Drug: bupivacaine; Device: Sham Adductor Canal Catheter

INTERVENTIONS:
Drug: ropivacaine — 15 ml 0.5% Ropivicaine for primary adductor canal block under ultrasound guidance and 0.2% Ropivicaine infusion 10 ml/hr.
  Other Names: Naropin
  Arms: Adductor Canal Catheter
Drug: bupivacaine — 20 ml bupivacaine ( Marcaine 0.25% with epinephrine 1:200000, Hospira Inc. Lake Forest, IL) diluted with 40 ml of normal saline injected intraoperatively into the knee joint before closure.
  Other Names: Marcaine
  Arms: Local Infiltration of Analgesia
Device: Sham Adductor Canal Catheter — Sham catheter placement via ultrasound-guided adductor canal block and 10ml/hr saline via OnQ Pump via continuous catheter in adductor canal.
  Arms: Local Infiltration of Analgesia
Device: Adductor Canal Catheter — Catheter placed in adductor canal via ultrasound guidance and continuous infusion via OnQ pump.
  Arms: Adductor Canal Catheter

SUMMARY:
The study is a prospective randomized controlled trial comparing local infiltration of analgesia in the knee joint and adductor canal catheters for postoperative analgesia following a primary Total Knee Arthroplasty (TKA).

DETAILED DESCRIPTION:
The study is a prospective, randomized controlled clinical trial comparing two methods of postoperative analgesia following primary TKA. Eligible primary TKA patients must be ASA I - III and require less than 20 mg oxycodone daily (or its equivalent). Exclusion criteria are: allergy to anesthetics, contraindication to regional anesthesia, sensory/ motor disorder involving operative limb, non-english speaking, ASA IV or greater, psychiatric or cognitive disorders, incarceration, renal insufficiency with Cr > 2.0 and hepatic failure. When patients agree to participate in the study the following data will be collected by the research staff: ASA physical status, age, height, weight, gender, quantitative opiate use, numeric pain score with visual descriptors, painDETECT score, WOMAC score and baseline Pain Management Questionnaire. When designated through randomization, local infiltration of analgesia will be placed intraoperatively by the surgeons, per usual protocol and patients in the LIA group will receive sham adductor canal catheter. All ACC's for both study groups will be placed postoperatively in the PACU. Those collecting data will be blinded from identifying patients in the control group, as both groups will have ACC placed with same technique. Potential risks for each procedure, which will be explained to the patient, include: bleeding, local infection, local anesthetic toxicity in the form of seizure and cardiac arrest and neuropathy. The preceding are commonly listed though infrequent complications of both procedures. Continuous ultrasound will guide the placement of the ACC. All adductor canal catheters will remain in for 72 hours. Pt from LIA group will be discharged home with sham catheter with a saline infusion at 10 ml/hr via an ambulatory pump. Patients in ACC group will be discharged with continuous adductor canal catheter delivering ropivacaine 0.2% at 10 ml/hr via an ambulatory pump. Patients will be called daily for pain diary results. As well as at 6-8 weeks postoperatively to collect painDetect and WOMAC survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85
* American Society of Anesthesiologists (ASA) Physical Status (PS) 1-3. • Undergoing Unilateral, Primary, Total Knee Arthroplasty
* English as native language

Exclusion Criteria:

* Patient refusal
* History of opioid dependence
* Contraindication to peripheral nerve block • Pre-existing significant neuropathy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain via numeric rating scale at rest and with activity during each physical therapy session | post-operative day #0 to post-operative day #3
  postoperative pain as measured by numeric rating scale at rest and with movement during each physical therapy session.

SECONDARY OUTCOMES:
Postoperative opioid consumption | post-operative day #0 to postoperative day # 3
  Opioid consumption during hospitalization in oxycodone equivalents at 24, 48 and 72 hours
Chronic post-surgical pain measured via validated painDetect and WOMAC questionnaires | 6-8 weeks after surgical date
  Assess post-surgical pain and function as measured by PainDetect and WOMAC questionnaires at 6-8 weeks post-operative compared to preoperative pain and function
Passive and Active Range of Motion during Physical Therapy | POD #0 to postoperative day #2
  Assess quantitative passive and active range of motion during physical therapy as well as Timed up to Go (TUG) which is routine assessment during physical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime L Baratta, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Background] Essving P, Axelsson K, Aberg E, Spannar H, Gupta A, Lundin A. Local infiltration analgesia versus intrathecal morphine for postoperative pain management after total knee arthroplasty: a randomized controlled trial. Anesth Analg. 2011 Oct;113(4):926-33. doi: 10.1213/ANE.0b013e3182288deb. Epub 2011 Aug 4. PMID 21821506
- [Background] Charous MT, Madison SJ, Suresh PJ, Sandhu NS, Loland VJ, Mariano ER, Donohue MC, Dutton PH, Ferguson EJ, Ilfeld BM. Continuous femoral nerve blocks: varying local anesthetic delivery method (bolus versus basal) to minimize quadriceps motor block while maintaining sensory block. Anesthesiology. 2011 Oct;115(4):774-81. doi: 10.1097/ALN.0b013e3182124dc6. PMID 21394001
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Kazak Bengisun Z, Aysu Salviz E, Darcin K, Suer H, Ates Y. Intraarticular levobupivacaine or bupivacaine administration decreases pain scores and provides a better recovery after total knee arthroplasty. J Anesth. 2010 Oct;24(5):694-9. doi: 10.1007/s00540-010-0970-x. Epub 2010 Jun 23. PMID 20571832